CLINICAL TRIAL: NCT07349238
Title: The Relationship Between Thoracic Kyphosis Angle and Shoulder Pain, Range of Motion, Isokinetic Muscle Strength, and Functionality
Brief Title: The Relationship Between Thoracic Kyphosis Angle and Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Assoc.Prof.Dr., Uskudar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Uskudar81
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Pain; Thoracic Kyphosis
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thoracic Kyphosis (Other): The group of participants to be evaluated
  Interventions: Other: Thoracic Kyphosis isokinetic measurement

INTERVENTIONS:
Other: Thoracic Kyphosis isokinetic measurement — Thoracic kyphotic angle was assessed by manual The group of participants to be evaluated, shoulder pain severity by Visual Analog Scale, shoulder range of motion by manual goniometer, shoulder isokinetic strength by isokinetic dynamometer, and upper extremity functionality by Quick Disability of the Arm, Shoulder, and Hand questionnaire.

SUMMARY:
This study aimed to investigate the correlation between increased thoracic kyphosis and these factors.

DETAILED DESCRIPTION:
Thoracic kyphosis angle was assessed with a manual inclinometer, shoulder pain severity with a Visual Analog Scale, shoulder range of motion with a manual goniometer, shoulder isokinetic strength with an isokinetic dynamometer, and upper extremity function with the Quick Disability of the Arm, Shoulder, and Hand questionnaire.

ELIGIBILITY:
Inclusion criteria:

* Being between 18 and 60 years of age,
* Having a thoracic kyphosis angle greater than 40°,
* Voluntary participation in the study.

Exclusion criteria:

* Having a diagnosis of neuromuscular disorder of the spine and upper extremities,
* Having received treatment for any spinal cord or upper extremity pathology in the last year,
* Systemic diseases or connective tissue disorders,
* Being pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the angle of thoracic kyphosis | 1 week
  Participants' thoracic kyphosis angle was assessed using two gravity-dependent manual inclinometers (Isomed Inc. 975 Sandy Blvd, Portland, USA). The manual inclinometer is a valid and reliable method used to measure range of motion and postural curvatures of the spine. During the measurement process, the feet of the inclinometers were positioned on the spinal protrusions that were identified as corresponding to the first and second thoracic vertebrae (T1/2) and the twelfth thoracic and first lumbar vertebrae (T12/L1). Spinal levels were determined through palpation while the subjects were in a natural standing position.
Visual Analog Scale | 1 week
  Participants' pain intensity was evaluated with the Visual Analog Scale , which consists of a 100 mm long, fixed horizontal line.Visual Analog Scale is considered one of the best available methods that are valid and reliable for estimating pain intensity. Participants were asked to mark the point representing the severity of shoulder pain in their current situation. The Visual Analog Scale score was determined by measuring the end of the line from the left beginning to the point marked by the patient, in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Yağmur Yarayan, Study Chair — Uskudar University
Locations (1):
- Sportomed Physical Therapy and Rehabilitation Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roghani T, Zavieh MK, Manshadi FD, King N, Katzman W. Age-related hyperkyphosis: update of its potential causes and clinical impacts-narrative review. Aging Clin Exp Res. 2017 Aug;29(4):567-577. doi: 10.1007/s40520-016-0617-3. Epub 2016 Aug 18. PMID 27538834
- [Background] Katzman WB, Wanek L, Shepherd JA, Sellmeyer DE. Age-related hyperkyphosis: its causes, consequences, and management. J Orthop Sports Phys Ther. 2010 Jun;40(6):352-60. doi: 10.2519/jospt.2010.3099. PMID 20511692
- [Background] Lewis JS, Valentine RE. Clinical measurement of the thoracic kyphosis. A study of the intra-rater reliability in subjects with and without shoulder pain. BMC Musculoskelet Disord. 2010 Mar 1;11:39. doi: 10.1186/1471-2474-11-39. PMID 20193055